CLINICAL TRIAL: NCT05964751
Title: the Association Between Metabolic Syndrome and Its Components With Lupus Nephritis in Systemic Lupus Erythematosus Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Salah Eldin Ali, resident at rheumatology and rehabilitation department, Sohag University
Other Study IDs: soh-Med-23-07-15MS
Record Dates: First submitted 2023-07-18; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patinets with lupus nephritis: patients diagnosed as lupus nehpritis
  Interventions: Diagnostic Test: lipid profile; Diagnostic Test: fasting blood suger
- pathents without lupus nephritis: sle pathients not diagnosed as lupus nephritis
  Interventions: Diagnostic Test: lipid profile; Diagnostic Test: fasting blood suger
- controls: controls will be matched for sex, age, and level of schooling withot history of connective tissue disorders, systemic active disease and renal history
  Interventions: Diagnostic Test: lipid profile; Diagnostic Test: fasting blood suger

INTERVENTIONS:
Diagnostic Test: lipid profile — measuerments of lipid profile parameters to detect hyperlipidemia
Diagnostic Test: fasting blood suger — measurment of fasting blood suger to detect hyprerglicemia

SUMMARY:
Systemic lupus erythematosus (SLE) is a heterogeneous autoimmune disease that involve s many different organs and display a variable clinical course. The prevalence of SLE varies across gender, race/ethnicity, and geographic regions. SLE demonstrates a striking female predominance with a peak incidence of disease during the reproductive years. In adults, the female to male ratio is 10-15:1.

Clinical features in individual patients can be quite variable and range from mild joint and skin involvement to severe, life-threatening internal organ disease. Constitutional symptoms, rash, mucosal ulcers, inflammatory polyarthritis, photosensitivity, and serositis are the most common clinical features of the disease .

Major organ affection in SLE includes Neuropsychiatric involvement (cognitive impairment, depression, psychosis, seizures, stroke, demyelinating syndromes, peripheral neuropathy, etc.) and cardiopulmonary manifestations. Lupus nephritis is the most common of the potentially life-threatening manifestations .

Renal involvement is common in SLE and is a significant cause of morbidity and mortality. It is estimated that as many as 90% of patients with SLE will have pathologic evidence of renal involvement on biopsy, but clinically significant nephritis will develop in only 50%.

Lupus involvement in the kidney manifests as urinary findings (proteinuria, hematuria, pathologic casts) with or without a rise in serum creatinine. The specific criteria listed for renal involvement are a urine protein > 500 mg/dL or red blood cell casts, Lupus nephritis is often confirmed by kidney biopsy, with the results showing one or more of the classes of lupus nephritis.

The metabolic syndrome is a prevalent disorder which is defined by the presence of central obesity, dyslipidemia, hypertension, and disturbed glucose metabolism . It is known that Metabolic syndrome predisposes to cardiovascular disease (CVD) and consequently, to a rise in CVD morbidity and mortality. This syndrome plays a major role in the complex network of systemic pro-inflammatory and prothrombotic states involved in the development of CVD .

Compared with patients without Metabolic syndrome, SLE patients from the multinational, multiethnic Systemic Lupus Erythematosus International Collaborating Clinics (SLICC) cohort with the diagnosis of Metabolic syndrome were older, had a higher disease activity, an increased number of recent disease flares, and had accrued more organ damage . Mok et al report that Metabolic syndrome is significantly associated with new organ damage, vascular events, and mortality in patients with SLE .

ELIGIBILITY:
Inclusion Criteria:

* 1. Age less than 18 years . 2. Patient not able and willing to give written informed consent. 3. Patients with pregnancy, cancer and with viral infectious diseases. 4. Patients with other autoimmune diseases rather than SLE.

Exclusion Criteria:

* 1. Age less than 18 years . 2. Patient not able and willing to give written informed consent. 3. Patients with pregnancy, cancer and with viral infectious diseases. 4. Patients with other autoimmune diseases rather than SLE.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Age less than 18 years . Patient not able and willing to give written informed consent. Patients with pregnancy, cancer and with viral infectious diseases. Patients with other autoimmune diseases rather than SLE.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
lipid profile (triglycerides) | 1 year
  to detect triglycerides level as apart of diagnosis of metabolic syndrome
blood pressure measurement | 1 year
  to detect if patients is hypertinsive or not as apart of diagnosis of metaboic syndrome
fasting blood suger | 1 year
  measurment of fasting blood suger to detect hyperglycemia as apart of diagnosis of metaboic syndrome
body mass index | 1 year
  measurement of weight & height to detect body mass index as apart of diagnosis of metaboic syndrome
protein creatinine ratio | 1 year
  to measure amount of protein in urine as apart of lupus nephritis
anti nuclear antibody test by IF | 1 YEAR
  this test to diagnose patient as SLE

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Pons-Estel GJ, Alarcon GS, Scofield L, Reinlib L, Cooper GS. Understanding the epidemiology and progression of systemic lupus erythematosus. Semin Arthritis Rheum. 2010 Feb;39(4):257-68. doi: 10.1016/j.semarthrit.2008.10.007. Epub 2009 Jan 10. PMID 19136143
- [Background] Lim SS, Bayakly AR, Helmick CG, Gordon C, Easley KA, Drenkard C. The incidence and prevalence of systemic lupus erythematosus, 2002-2004: The Georgia Lupus Registry. Arthritis Rheumatol. 2014 Feb;66(2):357-68. doi: 10.1002/art.38239. PMID 24504808
- [Background] DUBOIS EL, TUFFANELLI DL. CLINICAL MANIFESTATIONS OF SYSTEMIC LUPUS ERYTHEMATOSUS. COMPUTER ANALYSIS OF 520 CASES. JAMA. 1964 Oct 12;190:104-11. doi: 10.1001/jama.1964.03070150014003. No abstract available. PMID 14184513
- [Background] Hahn BH, McMahon MA, Wilkinson A, Wallace WD, Daikh DI, Fitzgerald JD, Karpouzas GA, Merrill JT, Wallace DJ, Yazdany J, Ramsey-Goldman R, Singh K, Khalighi M, Choi SI, Gogia M, Kafaja S, Kamgar M, Lau C, Martin WJ, Parikh S, Peng J, Rastogi A, Chen W, Grossman JM; American College of Rheumatology. American College of Rheumatology guidelines for screening, treatment, and management of lupus nephritis. Arthritis Care Res (Hoboken). 2012 Jun;64(6):797-808. doi: 10.1002/acr.21664. No abstract available. PMID 22556106